CLINICAL TRIAL: NCT03248973
Title: Successful Treatment of Maternal Listeria Monocytogenes Bacteremia in the First Trimester of Pregnancy: a Case Report and Review of Literatures
Brief Title: Successful Treatment of Maternal Listeria Monocytogenes Bacteremia in the First Trimester
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: 106030-C
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Listeria Monocytogenes
MeSH Terms: interventions — Ampicillin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ampicillin Injection — Ampicillin injection 2 g q4h for 3 weeks

SUMMARY:
Successful Treatment of Maternal Listeria Monocytogenes Bacteremia in the First Trimester of Pregnancy

DETAILED DESCRIPTION:
A 34-year-old nulliparous woman with 11 gestational weeks with flu-like illness was proved to be infection by Listeria monocytogenes, and then treated by intravenous ampicillin 2 g every 4 hours for 3 weeks. A healthy unaffected male baby was delivered at 41 weeks' gestation.

ELIGIBILITY:
Inclusion Criteria:

* One pregnant woman with listeria monocytogenes bacteremia in the first trimester

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One pregnant woman with listeria monocytogenes bacteremia in the first trimester
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Successful treatment | 1 month after delivery
  A favorable outcome of maternal listeria infection in the first trimester may be anticipated. Besides, intravenous ampicillin with or without gentamicin should be a reasonable treatment option for maternal listeria infection in the first trimester.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan